CLINICAL TRIAL: NCT05428865
Title: Correlation Between Body Mass Index, Selective Motor Control, Spasticity and Functional Ability in Children With Diplegic Cerebral Palsy
Brief Title: Correlation Between Body Mass Index, Selective Motor Control and Functional Ability in Children With CP
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Alaa Fahmy Hassan Al Nemr, PHD, Cairo University
Other Study IDs: P.T.REC/012/003833
Record Dates: First submitted 2022-06-11; First posted 2022-06-23 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Diplegic Cerebral Palsy
Keywords: isolated motor control; functional ability; body mass index; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: correlation study — investigate the correlations between body mass index, spasticity, functional ability and isolated motor control in children with spastic diplegia.

SUMMARY:
PURPOSE:

To investigate the correlations between body mass index, spasticity, functional ability and isolated motor control in children with spastic diplegia.

BACKGROUND:

Cerebral palsy is primarily a disorder of movement and posture

HYPOTHESES:

There is no correlation between body mass index, spasticity, functional ability and isolated motor control in children with spastic diplegia.

RESEARCH QUESTION:

Is there a correlation between body mass index, spasticity, functional ability and isolated motor control in children with spastic diplegia?

DETAILED DESCRIPTION:
This is an observational correlational study. SCALE will be used to assess selective motor control of lower extremity. GMFM-88 and WEE FIM will be used to assess functional ability. MAS will be used to assess degree of spasticity

ELIGIBILITY:
Inclusion Criteria:

* spastic diplegic CP, age from 6 to 9 years, able to follow verbal commands or instructions during testing procedures, 1+ and 2 according to Modified Ashworth scale (MAS), (GMFCS E&R) selected Level II , III.

Exclusion Criteria:

* patients who had contractures or fixed deformities related to the joints of the lower limbs, injection with Botulinium toxin or any orthopaedic surgery in lower limbs within one year before study,

Ages: 6 Years to 9 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: spastic diplegic cerebral palsy children
Sampling Method: Probability Sample
Enrollment: 84 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-07-24 (Actual)

PRIMARY OUTCOMES:
The selective control assessment of lower extremity (SCALE) | through study completion, an average of 1 year
  is a tool used for assessment of SVMC in children with spastic CP.
Anthropometric measurements | through study completion, an average of 1 year
  include weight (measured using a calibrated digital scale and height (measured using Harpenden Stadiometer). Body mass index (BMI) was calculated as weight (kg)/height (m2). higher scores indicate obesity
Wee Functional Independence Measure (Wee-FIM) | through study completion, an average of 1 year
  is a tool used to assess activities of daily living (ADL) in children with cerebral palsy.

SECONDARY OUTCOMES:
Modified Ashworth Scale (MAS) | through study completion, an average of 1 year
  For grading degree of spasticity.
Gross Motor Function Classification System Expanded and Revised for CP children between 6th and 12th birthday: | through study completion, an average of 1 year
  The Gross Motor Function Classification System (GMFCS E&R) is a classification system that describes the level of gross motor function of CP children according to abilities and limitations

CONTACTS AND LOCATIONS:
Overall Officials: Faculty OP Therapy, lecturer, Principal Investigator — Cairo University
Locations (1):
- Faculty Of Physical Therapy, Cairo, Egypt